CLINICAL TRIAL: NCT01217086
Title: Randomized, Double-blind, Parallel-group, Phase 3 Study
Brief Title: Program evaLuating the Autoimmune Disease iNvEstigational Drug cT-p13 in RA Patients(PLANETRA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Celltrion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CT-P13 3.1
Record Dates: First submitted 2010-10-04; First posted 2010-10-08 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Infliximab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CT-P13 (Active Comparator)
  Interventions: Drug: Infliximab
- Remicade (Active Comparator)
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Infliximab — Infliximab 3mg/kg is going to be administered for both arm as a 2-hour infusion per dose.
  Other Names: remicade

SUMMARY:
This is the trial to see how our product is similar to remicade by comparing the results of blood samples when co-administered with methotrexate between 12.5 to 25 mg/week, oral or parenteral dose and folic acid in rheumatoid arthritis patients who are not receiving adequate response to methotrexate alone up to week 30.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with active rheumatoid arthritis
* at least 3 months of treatment with methotrexate

Exclusion Criteria:

* have allergies to infliximab
* serious infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 617 (Actual)
Dates: Start 2010-10; Primary Completion 2011-11 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
PK equivalence to remicade | PK sampling at week 30

SECONDARY OUTCOMES:
efficacy endpoint | up to week 54.
  -ACR criteria comparison with Baseline at Weeks 14,30,54
efficacy endpoint | Up to week 54.
  - Time to onset of ACR20 response
efficacy endpoint | Up to week 54.
  - Mean decrease in disease activity measured by DAS28 comparison with Baseline at week 30
efficacy endpoint | Up to week 54.
  - Proportion of patients with a good response, defined according to the EULAR response criteria
efficacy endpoint | Up to week 54.
  - ACR20 at weeks 14 and 54
efficacy endpoint | Up to week 54.
  - ACR50 and ACR70 at weeks 14, 30, and 54
efficacy endpoint | Up to week 54.
  - Hybrid ACR response at weeks 14, 30, and 54
efficacy endpoint | Up to week 54.
  - SDAI and CDAI at weeks 14, 30, and 54
efficacy endpoint | Up to week 54.
  - Joint damage progression at week 54
efficacy endpoint | Up to week 54.
  - SF-36 at weeks 14, 30, and 54
efficacy endpoint | Up to week 54.
  - Fatigue
efficacy endpoint | Up to week 54.
  - Number of patients requiring salvage retreatment at weeks 30 and 54

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hyun Yoo, Principal Investigator — Hanyang University
Locations (1):
- Hanyang University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Eser A, Reinisch W, Schreiber S, Ahmad T, Boulos S, Mould DR. Increased Induction Infliximab Clearance Predicts Early Antidrug Antibody Detection. J Clin Pharmacol. 2021 Feb;61(2):224-233. doi: 10.1002/jcph.1732. Epub 2020 Sep 9. PMID 32905628
- [Derived] Yoo DH, Racewicz A, Brzezicki J, Yatsyshyn R, Arteaga ET, Baranauskaite A, Abud-Mendoza C, Navarra S, Kadinov V, Sariego IG, Hong SS, Lee SY, Park W. A phase III randomized study to evaluate the efficacy and safety of CT-P13 compared with reference infliximab in patients with active rheumatoid arthritis: 54-week results from the PLANETRA study. Arthritis Res Ther. 2016 Apr 2;18:82. doi: 10.1186/s13075-016-0981-6. PMID 27038608
- [Derived] Yoo DH, Hrycaj P, Miranda P, Ramiterre E, Piotrowski M, Shevchuk S, Kovalenko V, Prodanovic N, Abello-Banfi M, Gutierrez-Urena S, Morales-Olazabal L, Tee M, Jimenez R, Zamani O, Lee SJ, Kim H, Park W, Muller-Ladner U. A randomised, double-blind, parallel-group study to demonstrate equivalence in efficacy and safety of CT-P13 compared with innovator infliximab when coadministered with methotrexate in patients with active rheumatoid arthritis: the PLANETRA study. Ann Rheum Dis. 2013 Oct;72(10):1613-20. doi: 10.1136/annrheumdis-2012-203090. Epub 2013 May 16. PMID 23687260